CLINICAL TRIAL: NCT05459922
Title: Adjunctive Wearable Bright Light Therapy for Patients With Opioid Use Disorder: A Pilot Study
Brief Title: Adjunctive Bright Light Therapy for Opioid Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Chung Jung Mun, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00015561
Record Dates: First submitted 2022-06-07; First posted 2022-07-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder; Sleep Disturbance
Keywords: opioid use disorder; bright light therapy; reward function; methadone
MeSH Terms: conditions — Opioid-Related Disorders; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bright light therapy group (Experimental): Participants will receive 30-minute morning bright light therapy for 2 weeks. Participants will start the therapy within a few minutes of their designated wake up time, which is determined by their average wake time from the baseline week of sleep assessment.
  Interventions: Device: Wearable bright light therapy device
- Dim light (placebo) group (Placebo Comparator): Participants will receive 30-minute dim light (placebo) therapy for 2 weeks. Participants will start the therapy within a few minutes of their designated wake up time, which is determined by their average wake time from the baseline week of sleep assessment.
  Interventions: Device: Wearable placebo light therapy device

INTERVENTIONS:
Device: Wearable bright light therapy device — Light treatment glasses (Re-timer®) will be used to deliver bright light therapy. This device is available commercially and allows participants to freely move around while receiving light from LEDs positioned below the eyes. Re-timer® can be worn over glasses and does not interfere with vision, reading, or computer work.
  Arms: Bright light therapy group
Device: Wearable placebo light therapy device — The placebo Re-timer® emits light intensity to a level that will not impact sleep and circadian timing and appears identical to the original Re-timer®.
  Arms: Dim light (placebo) group

SUMMARY:
Investigators propose to conduct a pilot single-blind, parallel arm, randomized placebo-controlled trial evaluating the feasibility, acceptability, and preliminary efficacy of bright light therapy on reward system functioning among patients undergoing medication-assisted treatment for opioid use disorder.

DETAILED DESCRIPTION:
Bright light therapy (BLT) is a simple, safe, and accessible intervention that can effectively ameliorates sleep disruptions, as well as circadian misalignment and depressive symptoms, and could potentially improve reward system function among patients with OUD. Beyond seasonal affective disorder, BLT has shown efficacy as an intervention for non-seasonal depression, and post-traumatic stress disorder, which all exhibit significant impairment of the dopaminergic reward system and poor sleep quality as key symptoms. Investigators propose to conduct a pilot single-blind, parallel arm, randomized placebo-controlled trial evaluating the feasibility, acceptability, and preliminary efficacy of BLT on reward system functioning among patients undergoing medication-assisted treatment for OUD. The present study will establish feasibility for a larger randomized-clinical trial proposal.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65
* ability to speak, write, and read in English
* past 2 weeks of insomnia as evidenced by Insomnia Severity Index (ISI) total score of ≥10
* enrolled in outpatient medication-assisted treatment for OUD (i.e., either methadone or buprenorphine treatment)
* been in medication-assisted treatment for at least 3 months
* at least one month of stable methadone or buprenorphine dose
* have a smartphone

Exclusion Criteria:

* lifetime history of bipolar disorder or mania
* current narcolepsy, sleep paralysis, or restless leg syndrome as assessed by medical history
* history of seizure disorders/epilepsy
* the STOP-Bang score for obstructive sleep apnea ≥ 5
* retinal pathology, history of eye surgery or taking photosensitizing medications (e.g., lithium, L-tryptophan)
* current regular use of melatonin
* have circumstances that would interfere with study participation (e.g., impending jail sentence)
* previous experience with bright light therapy
* working a night shift or traveling outside the Arizona time zone in the past month
* pregnant, trying to get pregnant, or breastfeeding
* currently wearing prescription glasses with blue-light protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2022-10-23 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility--drop-out rate | At 2 weeks post-treatment
  From enrollment to post-treatment assessment
Feasibility--adherence to intervention | At 2 weeks post-treatment
  The number of days bright light therapy was completed divided by the total number of treatment days
Acceptability of the intervention | At 2 weeks post-treatment
  It will be measured by the Global Satisfaction subscale in an adapted version of the Treatment Satisfaction Questionnaire for Medication. The scores are calculated for each of the subscales, which range from 0 to 100, with higher scores indicating higher patient satisfaction with the intervention.
Changes in reward learning | Baseline and 2 weeks post-treatment
  Probabilistic Reward Task will be used to assess reward learning
Changes in reward valuation | Baseline and 2 weeks post-treatment
  Delayed Discounting Task will be used to assess reward valuation
Changes in Opioid Craving | Daily for the 1 week at baseline and throughout the treatment period (up to 2 weeks)
  To assess daily opioid craving, participants will be asked to rate the degree to which they have an urge to use illicit opioids in the moment on a 0-100 Visual Analogue Scale, with 0 being "Not at All" and 100 being "Extremely." This will be assessed multiple times per day via ecological momentary assessments. The timing of administration will be pseudo-randomized, but will broadly cover morning, midday and evening. Higher scores indicate greater opioid craving.

SECONDARY OUTCOMES:
Total Sleep Time (TST) | Daily for the 1 week at baseline and throughout the treatment period (up to 2 weeks)
  TST is defined as the total number of minutes asleep between the time a participant goes to bed at night and the time a participant gets out of bed in the morning. Total Sleep Time will be derived from wrist-worn actigraphy.
Sleep Onset Latency (SOL) | Daily for the 1 week at baseline and throughout the treatment period (up to 2 weeks)
  SOL is defined as the duration of time from turning the light off to falling asleep. SOL will be derived from wrist-worn actigraphy.
Wake After Sleep Onset (WASO) | Daily for the 1 week at baseline and throughout the treatment period (up to 2 weeks)
  WASO is defined as the total number of minutes awake following sleep initiation and before participants get out of bed in the morning. WASO will be derived from wrist-worn actigraphy.
Sleep Efficiency (SE) | Daily for the 1 week at baseline and throughout the treatment period (up to 2 weeks)
  SE is defined as sleep latency plus wake after sleep onset, and is calculated as the number of sleep minutes divided by the number of minutes in bed multiplied by 100. SE will be derived from wrist-worn actigraphy.
Illicit Opioid Use Frequency | Daily for the 1 week at baseline and throughout the treatment period (up to 2 weeks)
  Illicit opioid use will be assessed multiple times per day via ecological momentary assessments. The timing of administration will be pseudo-randomized, but will broadly cover morning, midday and evening.
Negative Affect | Daily for the 1 week at baseline and throughout the treatment period (up to 2 weeks)
  To assess daily negative affect, participants will be asked to rate several adjectives that describe negative affect on a 5-point Likert scale, with 1 being "No" and 5 being "Extremely." Items are based upon the Positive and Negative Affect Schedule. Negative affect will be assessed multiple times per day via ecological momentary assessments. The timing of administration will be pseudo-randomized, but will broadly cover morning, midday and evening. Higher scores indicate greater negative affect.
Positive Affect | Daily for the 1 week at baseline and throughout the treatment period (up to 2 weeks)
  To assess daily positive affect, participants will be asked to rate several adjectives that describe positive affect on a 5-point Likert scale, with 1 being "No" and 5 being "Extremely." Items are based upon the Positive and Negative Affect Schedule. Positive affect will be assessed multiple times per day via ecological momentary assessments. The timing of administration will be pseudo-randomized, but will broadly cover morning, midday and evening. Higher scores indicate greater positive affect.

CONTACTS AND LOCATIONS:
Overall Officials: Chung Jung Mun, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No